CLINICAL TRIAL: NCT06209879
Title: Managing Dry Eye in Rheumatoid Arthritis Patients With Dual-Polymer Hydroxypropyl Guar-and Hyaluronic Acid Containing Lubricant Eye Drops
Brief Title: Dual-Polymer Hydroxypropyl Guar-and Hyaluronic Acid Lubricants in Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, CHI-CHIN-SUN, Professor, School of Medicine Chang Gung University Taoyuan, Taiwan ; Doctor, Department of Ophthalmology, Chang Gung Memorial Hospital, Keelung, Taiwan, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 73583109
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Dry Eye Syndromes
Keywords: dry eye disease; rheumatoid arthritis; ocular lubricants; hydroxypropyl guar; hyaluronic acid
MeSH Terms: conditions — Dry Eye Syndromes; Arthritis, Rheumatoid | interventions — Fluorometholone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyaluronic Acid/Hydroxypropyl Guar arm (Experimental): Systane Hydration® MD
  Interventions: Drug: SYSTANE™ Hydration Lubricant Eye Drops

INTERVENTIONS:
Drug: SYSTANE™ Hydration Lubricant Eye Drops — SYSTANE™ Hydration Lubricant Eye Drops (Hyaluronic Acid [HA] 0.15%; Polyethylene Glycol 400 0.4%; Propylene Glycol 0.3%)1-2 drops 4 times a day) and 0.1% FML (1-2 drops 3 times a day) in both eyes for 12 week
  Other Names: 0.1% FML

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of hydroxypropyl guar-and hyaluronic acid containing lubricant eye drops in rheumatoid arthritis patients . The main question it aims to answer is:

• whether adding hydroxypropyl guar-and hyaluronic acid containing lubricant eye drops to steroid-based dry eye therapy improves dry eye symptoms in rheumatoid arthritis patients after 1 month.

Participants with rheumatoid arthritis will be treat with SYSTANE™ Hydration Lubricant Eye Drops (1-2 drops 4 times a day) and 0.1% Fluorometholone (1-2 drops 3 times a day) in both eyes for 12 weeks

DETAILED DESCRIPTION:
This is a prospective, single-center study designed to assess the efficacy of adding SYSTANE™ Hydration Lubricant Eye Drops on dry eyes secondary to rheumatoid arthritis (RA) patients. This study will enroll 40 dry-eye RA participants to achieve 32 evaluable participants for analysis. There are 4 phases throughout the whole study, including the screening phase (Day -30 to -14 [Visit 1]), the wash-out phase (Day -14±3 days to Day 0), baseline (Day 0 [Visit 2]), and the follow-up phase (Days 28±7 to 84±7 days [Visits 3 to 5]).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients in any race, 18 years (inclusive) or older.
2. Participants with a confirmed diagnosis of stable RA, determined by a rheumatologist according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) criteria. The systemic conditions of the enrolled patients were well controlled by their rheumatologists during the study period.
3. Patients diagnosed with the dry eye disease (DED) by an ophthalmologist based on the Tear Film & Ocular Surface Society Dry Eye Workshop II (TFOS DEWS II) dry eye severity grading diagnostic scheme criteria.
4. At screening, dry eye associated-RA patients on a steroid-based therapy who are stable in dry eye severity but experience/complain of persistent dry eye symptoms.

   The results within the range of the following assessments will be defined as stable DED with persistent dry eye symptoms at the screening phase:
   1. CFS score (NEI scale) 1-12.
   2. OSDI score 13-50.
5. In addition, patients should fulfill the required range of the following assessments at Visit 2:

   1. OSDI 13-50 scores
   2. Non invasive TBUT 3-10 seconds
   3. Schirmer's test (without anesthesia) 3-10 mm in 5 minutes
   4. CFS (NEI scale) 1-12 scores
6. Patients instilled the same dry eye therapeutic regimen of steroid eye drops and/or artificial tears (but naïve to HA-containing eye drops) for at least 3 months before the screening phase.

Exclusion Criteria:

1. Any known allergy to any of the study medications, conjunctival allergy or infectious disease, history of ocular chemical or thermal burn, Stevens-Johnson syndrome (SJS) or ocular pemphigoid, eyelid or lacrimal disease, any ocular operation within 6 months, grat versus host disease, non-dry-eye ocular inflammation, trauma, or presence of uncontrolled systemic disease.
2. Patients who have a history of intraocular, lacrimal or ocular surface surgery other than cataract extraction.
3. Patients who received cataract extraction surgery within 6 months of screening or patients who are planning to receive eye surgery during the study period.
4. Patients who wear corneal contact lens, have history of other severe systemic diseases, or other conditions, in the Investigator's opinion, may preclude enrollment.
5. Patients who received poly-pharmacy treatment for the dry eye before enrollment: DED requires topical ophthalmic treatment other than artificial tears and steroids (i.e., exclude auto-serum drops, diquafosol, and cyclosporine eye drops).
6. Patients with ocular conditions other than DED requiring topical ophthalmic treatment.
7. Patients who had experienced anti-rheumatic medication change within 3 months before the screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Change from baseline to the first month.
  The OSDI score is a 12-item patient-reported outcomes questionnaire with an overall score ranging from 0 to 100 to assess ocular surface symptoms, and the subjects can be categorized as having a normal (0-12), mild (13-22), moderate (23-32), or severe (33-100) ocular surface disease based on their OSDI score.

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | Change from baseline to second and third month
  The OSDI score is a 12-item patient-reported outcomes questionnaire with an overall score ranging from 0 to 100 to assess ocular surface symptoms, and the subjects can be categorized as having a normal (0-12), mild (13-22), moderate (23-32), or severe (33-100) ocular surface disease based on their OSDI score.
Non-invasive tear break-up time (TBUT) | Change from baseline to second and third month
  TBUT is used to assess the tear film stability by recording the interval between the last blink and the first appearance of a dry spot. TBUT less than 10 sec suggests an abnormal tear film. While TBUT between 5 to 10 sec is considered marginal, TBUT less than 5 sec indicates dry eye.
Corneal fluorescein staining (CFS) scores using National Eye Institute scale | Change from baseline to second and third month
  The CFS will be evaluated by external eye photography using the National Eye Institute (NEI) staining grid in which a score of 0 (normal) to 3 (severe) will be assigned to each of the 5 corneal regions (nasal, central, temporal, superior, and inferior). The CFS score will range between 0 and 15, and the maximum score of 15 indicates severe epitheliopathy.
Schirmer's test scores | Change from baseline to second and third month
  Schirmer's test is a quantitative test to measure maximal tear secretion capacity. A filter paper will be placed in the lower fornix for 5 min and the and the length of wetted paper is measured.While a Schirmer's test score of greater than 10 mm/5 min is classified as normal, test score of less than 5 mm/5 min indicates tear deficiency.
Tear meniscus height | Change from baseline to second and third month
  Tear meniscus height is a quantitative test to measure vertical height of the marginal tear strip

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Chin Sun, M.D/Ph.D, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Keelung Chang Gung memorial hospital, Keelung, Taiwan